CLINICAL TRIAL: NCT00520390
Title: A Phase I, Multicenter, Open-Label, Dose-Escalation Study Evaluating the Safety and Tolerability of Intravenous EZN-2208 PEG-SN38) Administered Weekly for 3 Weeks in 4-Week Cycles in Patients With Advanced Solid Tumors or Ymphoma (EZN-2208-02)
Brief Title: A Phase I, Study to Evaluate the Safety and Tolerability of Intravenous EZN-2208 in Patients With Advanced Solid Tumors or Lymphoma (EZN-2208-02)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enzon Pharmaceuticals, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EZN-2208-02
Record Dates: First submitted 2007-08-23; First posted 2007-08-24 (Estimated); Last update posted 2010-04-02 (Estimated); Status verified 2010-04

CONDITIONS: Lymphoma; Advanced Solid Tumors
MeSH Terms: conditions — Lymphoma | interventions — EZN-2208

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: EZN-2208

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of EZN-2208 that can be given to patients with advanced cancer or lymphoma. The safety of the study drug and its effect on the disease will also be studied.

Enzon will also perform pharmacokinetic (PK) testing of EZN-2208. PK testing measures the amount of a drug in the body at different time points.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of advanced and/or metastatic solid tumor or lymphoma that is refractory to standard therapy
* Measurable or evaluable disease
* Score of 0 to 2 on the ECOG performance scale

Exclusion Criteria:

* Concurrent serious medical illness
* Known, clinically suspected, or history of central nervous system (CNS) tumor involvement
* Active diarrhea
* Known history of coagulation disorder
* Patients requiring cytochrome P450 3A4 (CYP3A4) enzyme inducing medications
* Requirement for ketoconazole or other strong inhibitor of CYP3A4 enzymes
* Prior chemotherapy, immunotherapy, investigational agent, or other therapy used to treat the cancer within 4 weeks (6 weeks for prior treatment with mitomycin C or nitrosoureas) prior to the scheduled administration of EZN-2208.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34
Dates: Start 2007-05

PRIMARY OUTCOMES:
Determine the MTD of i.v. EZN-2208 administered weekly for 3 weeks in a 4-week cycle and recommended Phase 2 dose of i.v. EZN-2208

SECONDARY OUTCOMES:
Evaluate the safety and tolerability of EZN-2208, assess the pharmacokinetic PK profile of EZN-2208, SN38, and SN38G. | 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Amita Patnaik, M.D., Principal Investigator — South Texas Accelerated Research Therapeutics
Locations (1):
- South Texas Accelerated Research Therapeutics, San Antonio, Texas, United States

REFERENCES:
- [Derived] Park EJ, Choi J, Lee KC, Na DH. Emerging PEGylated non-biologic drugs. Expert Opin Emerg Drugs. 2019 Jun;24(2):107-119. doi: 10.1080/14728214.2019.1604684. Epub 2019 Apr 19. PMID 30957581